CLINICAL TRIAL: NCT03057665
Title: Atomic Magnetometer for Fetal Biomagnetism
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: H-2008-0099
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Fetal Heart Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant Women: Measure magnetic field versus time for fetus, using atomic biomagnetometer.
  Interventions: Device: Atomic Biomagnetometer

INTERVENTIONS:
Device: Atomic Biomagnetometer — Measure magnetic field of fetal heartbeat

SUMMARY:
The goal of this study is the evaluation of an atomic magnetometer that is practical for human biomagnetism studies. The investigators have built a device that has the necessary sensitivity, and will be testing it on a small number of adults and approximately 30 healthy pregnant subjects, in preparation for beginning pre-clinical studies of high-risk pregnancies.

DETAILED DESCRIPTION:
The goal of this study is evaluation of our atomic magnetometer for adult and fetal MCG studies. The investigators will assess the signal-to-noise and bandwidth performance under human acquisition conditions. They will also gain experience with the practical issues associated with making the measurements on human subjects.

The measurement sessions will take place in the magnetically shielded room in the UW Biomagnetism Laboratory, where similar studies have been made with SQUID detectors for more than 20 years, without incident. The room contains a bed and/or chair on which the subject may comfortably lie or sit.

The subject will remove all metal and magnetic objects (e.g. watches, glasses, jewelry, coins) and change into metal-free clothing. The subject will put on laser eye protection goggles. The subject will lie or sit on the patient bed in the magnetically shielded room with his or her chest (or stomach in the case of a pregnant mother) as close as possible to the magnetometer (typically 1 cm away), and will be monitored closely through a small opening in the shielded room to ensure comfort throughout the study. Positioning of the device with respect to the patient will be done by one of the researchers. In the case of pregnant women, an ultrasound will be taken to ascertain the position of the baby and facilitate initial positioning of the magnetometer. Depending on need for possible further positioning, the researcher may or may not leave the room after device positioning. The subject will be asked to remain still during data acquisition. (Should the subject become uncomfortable or simply need to move around, he or she will have complete freedom to do so and that particular measurement will be terminated.) Visual and audio contact with the subject will be maintained at all times via an open window in the magnetically shielded room. Using the atomic magnetometer, up to five-minute MCG recordings will be made at several locations in order to map the signal. The recordings will be analyzed off-line. An MCG or fMCG may also be recorded with Dr. Wakai's commercial Magnes and Tristan SQUID magnetometers, using similar acquisition parameters and processing procedures as for the AM. The purpose of the SQUID measurement is to compare the attained waveforms. Processing procedures for the SQUID data are identical to the atomic magnetometer data.

A typical recording session will consist of about 10 minutes for magnetometer alignment and optimization, followed by several 5-minute magnetometer acquisition periods separated by rest breaks during which the subject can relax and preliminary data analysis will be conducted by the researchers. The session may be completed by a SQUID measurement, requiring an additional 15 minutes, and by a brief exit interview to see if the subject had any comfort issues that were not identified during the session. The total recording session will take up to 2 hours .

ELIGIBILITY:
Inclusion Criteria:

* The subjects will be asked if they consider themselves healthy, if they are able to sit or lie still for 5 minute periods during data acquisition, if they have large metal plates, screws, or devices, and if they are pregnant.

Exclusion Criteria:

* Participants who self-identify as being unhealthy or having complications with their pregnancy. In addition, vulnerable populations such as prisoners, veterans, individuals with impaired decision-making capabilities, and non-English speakers will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 35 normal, nominally healthy adult volunteers (18 years or older) will be studied, including 30 pregnant women. The pregnant women will be healthy women with uncomplicated pregnancies. They will be studied at gestational ages 18-38 weeks, with studies terminating at 38 weeks or before. The non-pregnant adults will be either the PIs or other volunteers who do not have status relationship to the study investigators.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Atomic Magnetometer | 20-35 week gestation period
  Measure single-to-noise for acquisition of fetal magnetocardiograms

CONTACTS AND LOCATIONS:
Overall Officials: Thad Walker, PhD, Principal Investigator — Univ. of Wisconsin-Madison
Locations (1):
- Biomagnetism Laboratory, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No